CLINICAL TRIAL: NCT00838019
Title: Pilot Study About Viability and Efficacy of Intrabone Administration of Umbilical Cord Blood for Allogeneic Stem Cell Transplantation
Brief Title: Intrabone Cord Blood Transplantation
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Dr. Raimundo Belenes, Chief Executive Officer, Hospital Clinic.University of Barcelona
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TPH/SCU-IMed 01/08
Record Dates: First submitted 2009-02-05; First posted 2009-02-06 (Estimated); Last update posted 2009-02-06 (Estimated); Status verified 2009-02

CONDITIONS: Hematological Malignancies
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cord blood (Experimental)
  Interventions: Procedure: Intrabone administration of umbilical cord blood

INTERVENTIONS:
Procedure: Intrabone administration of umbilical cord blood — Single administration

SUMMARY:
The purpose of this study is to evaluate the viability of intrabone administration of umbilical cord blood as allogenic transplantation for the treatment of hematologic malignancies.

ELIGIBILITY:
Inclusion Criteria:

* Hematological malignancies
* Indication of allogenic transplantation
* No suitable donor (related/unrelated)
* No suitable cord blood unit with enough cellularity for standard transplant
* Written informed consent

Exclusion Criteria:

* ECOG > 2
* Co-morbidities
* HIV positive serology
* Pregnancy or breastfeeding
* Psychiatric illness

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2009-02; Primary Completion 2011-02 (Estimated); Study Completion 2011-02 (Estimated)

PRIMARY OUTCOMES:
Kinetics of hematopoietic engraftment | days 14, 21, 28 after administration

SECONDARY OUTCOMES:
Dynamics and chimerism of hematological engraftment | days 14, 21, 28 after administration

CONTACTS AND LOCATIONS:
Overall Officials: Montserrat Rovira, MD, Principal Investigator — Hospital Clinic of Barcelona
Locations (1):
- BMT Unit Hematology Department Hospital Clinic, Barcelona, Barcelona, Spain